CLINICAL TRIAL: NCT03174470
Title: Safety Demonstration of Increasing Intensities of Electrical Stimulation Delivered to The Bulbospongiosus Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virility Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VM-Rev-001
Record Dates: First submitted 2017-05-28; First posted 2017-06-02 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENS stimulator (Experimental): Single day Transcutaneous electrical nerve stimulations utilizing a commercial TENS stimulator (TensMed S82 ENRAF-NONIUS)
  Interventions: Device: TENS Stimulator

INTERVENTIONS:
Device: TENS Stimulator — Initial stimulation of arm (conditioning) followed by Increasing Intensities of Electrical Stimulation Delivered to The Bulbospongiosus Muscle
  Other Names: TensMed S82 ENRAF-NONIUS

SUMMARY:
The company suggests a new concept of treatment for PE: Transient inhibition of striated muscle contraction by a transcutaneous stimulation device. This study aim is to evaluate the safety of delivering increasing electrical stimulation intensities to the subject's perineum, using a TENS technique and equipment, followed by a 72-hour postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Ability to follow study instructions and complete study assessment tools

Exclusion Criteria:

* History of cardiovascular disorders
* Any type of implanted pacemaker/defibrillator
* Hypertension
* Diabetes Mellitus
* Local dermatological disease
* Local skin irritation/lesions
* Any neurological disorder
* Any psychiatric disease and/or psychiatric medications

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline
  Pain sensation score given by all subjects, as well as their verbal description of what they sensed during the various stimulations

SECONDARY OUTCOMES:
Incidence of post-treatment Adverse Events | 72 hours
  Post treatment safety evaluation completed by subjects (using safety questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No